CLINICAL TRIAL: NCT06887504
Title: The Evaluation of White Matter Intensities in Patients with Pediatric Epilepsy
Status: Completed | Type: Observational
Sponsor: Aysen Orman (Other)
Responsible Party: Sponsor-Investigator, Aysen Orman, Associate Prof, Mersin University
Organization: Mersin University (Other)
Other Study IDs: Balikesir Univercity
Record Dates: First submitted 2025-02-17; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Epilepsies; White Matter Alterations
Keywords: Children; epilepsy; white matter; hyperintensity
MeSH Terms: conditions — Epilepsy; Leukoaraiosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients diagnosed with epilepsy who underwent epilepsy protocol cranial MRI between 01.08.2019 and: All patients underwent imaging on a 1.5 T MRI device (Ingenia, release 5.3-5.7 software, Philips Medical Systems, Best, the Netherlands). The epilepsy protocol consisted of axial T1-weighted imaging (WI) spin-echo (SE)(repetition time/echo time (TR/TE): 450/15; field of view (FOV): 230 mm, slice thickness: 5 mm, matrix: 308 ×183), axial fat suppressed (FS) T1-WI SE(TR/TE: 633/15; field of view (FOV): 230 mm, slice thickness: 5 mm, matrix: 308 × 183), axial T2-WI turbo spin-echo (TSE) (TR/TE: 5240/100, FOV: 230 mm, slice thickness: 5 mm, matrix: 384 × 237), coronal FS fluid- attenuated inversion recovery (FLAIR) sequence (TR/TE: 11,000/130; FOV: 230 mm, slice thickness: 5 mm, matrix: 256 × 157), coronal T2-WI TSE (TR/TE: 3027/100; FO): 200 mm, slice thickness: 3 mm, matrix: 336 × 217), coronal T1-WI inversion recovery (IR) (TR/TE: 3079/15; field of view (FOV): 200 mm, slice thickness: 3.5 mm, matrix: 336 × 211), coronal FLAIR sequence (TR/TE: 11,000/130; FOV: 230 mm, slice thic

SUMMARY:
Aim: Neuroimaging is an important tool, in combination with a detailed medical history, physical examination, and electroencephalography, in the diagnosis and classification of epilepsy. White matter hyperintensities (WMHs) are bright areas of high signal intensity seen in white matter at T2-weighted MRI. Researchers aimed to evaluate whether white matter hyperintensities are more common in children with epilepsy.

Material-method: Patients who underwent cranial MRI with diagnoses of epilepsy based on International League Against Epilepsy (ILAE) criteria at the Balıkesir University Medical Faculty Pediatric neurology clinic, Türkiye, between 01.08.2019 and 01.03.2024 and patients who underwent cranial MRI during the same period due to indications other than epilepsy, such as headache, syncope, and vertigo, were included in the study. Written informed consent was received from all patients.

DETAILED DESCRIPTION:
Aim: Neuroimaging is an important tool, in combination with a detailed medical history, physical examination, and electroencephalography, in the diagnosis and classification of epilepsy. White matter hyperintensities (WMHs) are bright areas of high signal intensity seen in white matter at T2-weighted MRI. Researchers aimed to evaluate whether white matter hyperintensities are more common in children with epilepsy.

Material-method: Patients who underwent cranial MRI with diagnoses of epilepsy based on International League Against Epilepsy (ILAE) criteria at the Balıkesir University Medical Faculty Pediatric neurology clinic, Türkiye, between 01.08.2019 and 01.03.2024 and patients who underwent cranial MRI during the same period due to indications other than epilepsy, such as headache, syncope, and vertigo, were included in the study. Written informed consent was received from all patients.

ELIGIBILITY:
Inclusion Criteria:

Cranial MRI during the same period due to indications other than epilepsy;

* headache
* syncope and
* vertigo

Exclusion Criteria:

Patients with neuropsychiatric disorders;

* depression,
* psychotic disorders,
* autism spectrum disorder History of medication use for any chronic disease other than seizure medication, History of vascular disease ;
* Collagen tissue diseases;
* lupus,
* juvenile rheumatoid arthritis,
* polyarteritis nodosa,
* Kawasaki disease Demyelinating disease
* acute demyelinating disease (ADEM),
* Multiple sclerosis Acute symptomatic seizure or a single unprovoked seizure, İncomplete file data, or MRI performed at a location other than our hospital

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male and Female
Study Population: The study group included patients diagnosed with epilepsy who underwent cranial MRI according to the epilepsy protocol between 01.08.2019 and 01.03.2024, and the control group included patients who underwent cranial MRI according to the standard protocol for indications other than epilepsy. Patients with psychiatric disorders, a history of any chronic disease other than seizure medication, a history of vascular disease or demyelinating disease, acute symptomatic seizures or a single unprovoked seizure, incomplete file data, and MRI performed at a location other than the hospital were excluded from the study. The age and weight of patients diagnosed with epilepsy, seizure type, anti-seizure medications used, and EEG findings were recorded retrospectively from the hospital information system module, and cranial MRI images were recorded retrospectively from the PACS archive system.
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
The Evaluation of White Matter Intensities in Patients with Pediatric Epilepsy | 01.08.2019 and 01.03.2024
  To determine whether white matter hyperintensities are more frequent in children with epilepsy by comparing epilepsy and control groups.
The Evaluation of White Matter Intensities in Patients with Pediatric Epilepsy | 01.08.2019 and 01.03.2024
  Better understanding the association between pediatric epilepsy patients and white matter changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol